CLINICAL TRIAL: NCT06305767
Title: A Phase 1/2 Study of V940 Plus Pembrolizumab With or Without Enfortumab Vedotin in Muscle-Invasive Urothelial Carcinoma (MIUC) (INTerpath-005)
Brief Title: A Clinical Study of Intismeran Autogene (V940) Treatment and Pembrolizumab in People With Bladder Cancer (V940-005/INTerpath-005)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V940-005; V940-005 (Other: MSD); U1111-1292-1952 (Registry Identifier: UTN); 2023-505658-17-00 (Registry Identifier: EU CT); INTerpath-005 (Other: MSD)
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enfortumab vedotin; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The Phase 2 Adjuvant Cohort is a placebo- and active-controlled, parallel-group, multicenter, double-blind safety and efficacy study of adjuvant intismeran autogene plus pembrolizumab versus adjuvant placebo plus pembrolizumab in participants with pathologic high-risk MIUC after radical resection. Eligible participants will be randomly assigned in a 1:1 ratio to receive treatment with either intismeran autogene plus pembrolizumab or placebo plus pembrolizumab.
  The Phase 1 Perioperative Cohort of this study has a single arm into which eligible participants are allocated. It will evaluate safety and preliminary efficacy of perioperative (neoadjuvant and adjuvant) intismeran autogene in combination with pembrolizumab plus EV for participants with muscle-invasive bladder cancer (MIBC).
Who Masked: Participant, Investigator
Masking Description: The Phase 2 Adjuvant Cohort of study will be conducted as a double-blind study under in-house blinding procedures. Intismeran autogene and placebo will be prepared and dispensed by unblinded pharmacists and administered in a blinded fashion by blinded personnel. The participants and the investigators who are involved in the study intervention administration will be unaware of the intervention assignments.
  The Phase 1 Perioperative Cohort will be conducted as an open-label study. Participants and investigators will be aware of the intervention assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Adjuvant Cohort: Pembrolizumab + Intismeran autogene (Experimental): Adjuvant Cohort participants receive adjuvant treatment with up to 9 cycles of pembrolizumab plus up to a total of 9 doses of intismeran autogene. Intismeran autogene doses may begin as soon as Day 22 of Cycle 1. The total duration of treatment is up to approximately 13 months.
  Interventions: Biological: Pembrolizumab; Biological: Intismeran autogene
- Adjuvant Cohort: Pembrolizumab + Placebo (Active Comparator): Adjuvant Cohort participants receive adjuvant treatment with up to 9 cycles of pembrolizumab plus up to a total of 9 doses of placebo. Placebo doses may begin as soon as Day 22 of Cycle 1. The total duration of treatment is up to approximately 13 months.
  Interventions: Biological: Pembrolizumab; Other: Placebo
- Perioperative Cohort: Pembrolizumab + Intismeran autogene + EV and Surgery (Experimental): Participants will receive neoadjuvant treatment with up to 4 cycles of pembrolizumab plus EV and 1 to 4 doses of intismeran autogene, followed by radical cystectomy [RC] plus pelvic lymph node dissection [PLND], and then adjuvant treatment with up to 13 cycles of pembrolizumab plus up to 5 cycles of EV and 5 to 8 doses of intismeran autogene (for a total of 9 neoadjuvant plus adjuvant Intismeran autogene doses), or until any of the protocol-specified criteria for discontinuation of study intervention are met. The total duration of treatment is up to approximately 16 months.
  Interventions: Biological: Pembrolizumab; Biological: Intismeran autogene; Biological: Enfortumab Vedotin; Procedure: Surgery (RC plus PLND)

INTERVENTIONS:
Biological: Pembrolizumab — Administered via intravenous (IV) infusion at a dose of 400 mg on Day 1 of every 6-week cycle for up to 9 adjuvant cycles for Adjuvant Cohort participants, or at a dose of 200 mg on Day 1 of every cycle for up to four 3-week neoadjuvant cycles and up to thirteen 3-week adjuvant cycles for Perioperative Cohort participants.
  Other Names: MK-3475; Keytruda®
Biological: Intismeran autogene — Administered via intramuscular (IM) injection at a dose of 1 mg every 3 weeks for a total of up to 9 adjuvant doses for Adjuvant Cohort participants, or at a dose of 1 mg every 3 weeks for a total of up to 9 doses in the neoadjuvant and adjuvant periods for Perioperative Cohort participants.
  Other Names: V940
  Arms: Adjuvant Cohort: Pembrolizumab + Intismeran autogene; Perioperative Cohort: Pembrolizumab + Intismeran autogene + EV and Surgery
Other: Placebo — Intismeran autogene diluent only (saline and/or dextrose) administered via IM injection Q3W for up to 9 doses.
  Arms: Adjuvant Cohort: Pembrolizumab + Placebo
Biological: Enfortumab Vedotin — Administered via IV infusion at a dose of 1.25 mg/kg on Day 1 and Day 8 of every cycle for up to four 3-week neoadjuvant cycles and up to five 3-week adjuvant cycles for Perioperative Cohort participants.
  Other Names: PADCEV®
  Arms: Perioperative Cohort: Pembrolizumab + Intismeran autogene + EV and Surgery
Procedure: Surgery (RC plus PLND) — Curative intent surgery (RC plus PLND) will be administered to all participants in the Perioperative Cohort and will be done in accordance with the American Urological Association/American Society for Radiation Oncology/American Society of Clinical Oncology/Society of Urologic Oncology guidelines. RC plus PLND will be performed within 6 weeks of the last dose of neoadjuvant intismeran autogene plus pembrolizumab plus EV treatment. Adjuvant intismeran autogene plus pembrolizumab plus EV treatment will begin within 8 weeks of completing RC plus PLND.
  Arms: Perioperative Cohort: Pembrolizumab + Intismeran autogene + EV and Surgery

SUMMARY:
Researchers are looking for new ways to treat people with high-risk muscle-invasive urothelial carcinoma (MIUC). Urothelial carcinoma is a type of bladder cancer that begins in cells that line the inside of the bladder and other parts of the urinary tract, such as part of the kidneys, ureters, and urethra. People with MIUC usually have chemotherapy before surgery, then surgery to remove the cancer. Chemotherapy is a type of medicine to destroy cancer cells or stop them from growing. After surgery, some people receive more treatment to prevent cancer from returning. Pembrolizumab is an immunotherapy, which is a treatment that helps the immune system fight cancer. Enfortumab vedotin (EV) is an antibody drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells. Researchers want to learn if giving intismeran autogene (the study treatment) with pembrolizumab can prevent MIUC from returning after surgery. Intismeran autogene (also called mRNA-4157) is designed to treat each person's cancer by helping the person's immune system identify and kill cancer cells based on certain proteins found on those cancer cells.

The goals of this study are to learn if people who receive intismeran autogene and pembrolizumab are alive and cancer free longer than those who receive placebo and pembrolizumab, and to learn about the safety of intismeran autogene, pembrolizumab, and EV, and if people tolerate them.

DETAILED DESCRIPTION:
Enrollment of participants into the Phase 1 Perioperative Cohort of this study is planned to start in approximately April of 2025.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a histological diagnosis of urothelial carcinoma (UC)
* Must provide blood samples per protocol, to enable intismeran autogene production, and circulating tumor deoxyribonucleic acid testing
* Has an Eastern Cooperative Oncology Group performance status of 0 to 2 assessed within 7 days before randomization
* Must provide a formalin-fixed paraffin-embedded tumor tissue sample for next generation sequencing

Adjuvant Cohort:

* Has MIUC
* Has high-risk pathologic disease after radical resection
* For participants who have not received cisplatin-based neoadjuvant chemotherapy, are ineligible to receive cisplatin according to protocol pre-defined criteria

Perioperative Cohort:

* Has MIBC
* Is deemed eligible for RC and PLND and agrees to undergo curative intent standard RC and PLND and neoadjuvant and adjuvant treatment per protocol
* Is ineligible to receive cisplatin according to protocol pre-defined criteria

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has known additional malignancy that is progressing or has required active treatment ≤3 years prior to study randomization
* Has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has active hepatitis B and hepatitis C virus infection

Adjuvant Cohort:

* Has received prior systemic anticancer therapy
* Has received prior neoadjuvant therapy, with the exception of neoadjuvant cisplatin-based chemotherapy for MIUC
* Has severe hypersensitivity to either intismeran autogene or pembrolizumab (MK-3475) and/or any of their excipients

Perioperative Cohort:

* Has received any prior systemic treatment, cancer vaccine treatment, chemoradiation, and/or radiation therapy treatment for MIBC
* Has severe hypersensitivity to either intismeran autogene, pembrolizumab, or EV and/or any of their excipients
* Has ongoing sensory or motor neuropathy
* Has active keratitis or corneal ulcerations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2031-10-20 (Estimated)

PRIMARY OUTCOMES:
Adjuvant Cohort: Disease Free Survival (DFS) | Up to approximately 28 months
  DFS is defined as the time from randomization until death from any cause, or presence of disease per investigator assessment with muscle-invasive (≥pT2) disease or any high-grade non-muscle invasive disease in the urothelial tract (upper tract or lower tract) on imaging and biopsy, and/or disease recurrence outside the urothelial tract on imaging with or without confirmation by biopsy. DFS will be reported for the Adjuvant Cohort.
Perioperative Cohort: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 19 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience AEs will be reported for the Perioperative Cohort.
Perioperative Cohort: Number of Participants Who Discontinue Study Treatment Due to AE | Up to approximately 16 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinue study treatment due to an AE will be reported for the Perioperative Cohort.

SECONDARY OUTCOMES:
Adjuvant Cohort: Overall Survival (OS) | Up to approximately 28 months
  Overall survival is defined as the time from randomization to death due to any cause. OS will be reported for the Adjuvant Cohort.
Adjuvant Cohort: Distant Metastasis-Free Survival (DMFS) | Up to approximately 28 months
  DMFS is defined as the time from randomization until death from any cause, or disease recurrence outside the urothelial tract on imaging with or without confirmation by biopsy, per investigator assessment. DMFS will be reported for the Adjuvant Cohort.
Adjuvant Cohort: Number of Participants Who Experience an AE | Up to approximately 16 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who experience an AE will be reported for the Adjuvant Cohort.
Adjuvant Cohort: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 13 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of participants who discontinue study treatment due to an AE will be presented for the Adjuvant Cohort.
Perioperative Cohort: Pathologic Complete Response (pCR) Rate | Up to approximately 18 weeks
  pCR is defined as the absence of viable tumor (pT0N0) in examined tissue from RC plus PLND as assessed by the investigator. pCR rate will be reported as the percentage of participants in the Perioperative Cohort having pCR.
Perioperative Cohort: Pathologic Downstaging (pDS) Rate | Up to approximately 18 weeks
  pDS is defined as participants with <pT2 (includes pT0, pTis, pTa, pT1) and N0 in examined tissue from RC plus PLND as assessed by the investigator. pDS rate will be reported as the percentage of participants in the Perioperative Cohort having pDS.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (74):
- United States (10):
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 140)-Department of Urology/Institute of Uro ( Site 0104), Los Angeles, California
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlandoc ( Site 0102), Orlando, Florida
  - University of Chicago Medical Center ( Site 0109), Chicago, Illinois
  - University of Iowa ( Site 0110), Iowa City, Iowa
  - Icahn School of Medicine at Mount Sinai ( Site 0101), New York, New York
  - Duke Cancer Institute ( Site 0107), Durham, North Carolina
  - Cleveland Clinic Main ( Site 0100), Cleveland, Ohio
  - Fox Chase Cancer Center ( Site 0106), Philadelphia, Pennsylvania
  - UT Southwestern Medical Center ( Site 0103), Dallas, Texas
  - Houston Methodist Hospital-Department of Urology ( Site 0111), Houston, Texas
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 1803), Macquarie University, New South Wales
  - Westmead Hospital ( Site 1802), Westmead, New South Wales
  - Mater Misericordiae Limited ( Site 1808), South Brisbane, Queensland
  - One Clinical Research ( Site 1807), Nedlands, Western Australia
- Canada (5):
  - BC Cancer Vancouver ( Site 0004), Vancouver, British Columbia
  - Princess Margaret Cancer Centre ( Site 0003), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0005), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0001), Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer ( Site 0002), Sherbrooke, Quebec
- Chile (5):
  - Bradfordhill-Clinical Area ( Site 1501), Recoleta, Santiago, Region M. de Santiago
  - FALP ( Site 1500), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1503), Santiago, Region M. de Santiago
  - CIDO SpA ( Site 1509), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 1506), Viña del Mar, Región de Valparaíso
- Colombia (4):
  - Clínica Universitaria Colombia ( Site 1600), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 1605), Valledupar, Cesar Department
  - Instituto Nacional De Cancerologia-Oncología Clínica ( Site 1606), Bogota, Cundinamarca
  - Fundacion Valle del Lili- CIC-Oncology CIC ( Site 1608), Cali, Valle del Cauca Department
- France (5):
  - Oncopole Claudius Regaud ( Site 0302), Toulouse, Haute-Garonne
  - Institut de Cancérologie de l'Ouest ( Site 0300), Angers, Maine-et-Loire
  - Hopital Claude Huriez - CHU de Lille ( Site 0301), Lille, Nord
  - Hôpital Saint-Louis ( Site 0304), Paris
  - Gustave Roussy ( Site 0303), Villejuif, Île-de-France Region
- Germany (5):
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Site 0401), Munich, Bavaria
  - Caritas-Krankenhaus St. Josef-Klinik fuer Urologie ( Site 0404), Regensburg, Bavaria
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Urologie ( Site 0405), Dresden, Saxony
  - Universitätsklinikum Halle-Universitätsklinik und Poliklinik für Urologie ( Site 0402), Halle, Saxony-Anhalt
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0400), Berlin
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 0504), Rome, Lazio
  - Ospedale San Martino-U.O. Oncologia Medica 1 ( Site 0500), Genoa, Liguria
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0502), Milan, Lombardy
  - Azienda Ospedaliera Di Rilievo Nazionale A. Cardarelli-UOSC Oncologia ( Site 0503), Naples, Napoli
  - Ospedale San Raffaele-Oncologia Medica ( Site 0501), Milan
- Auckland City Hospital ( Site 1901), Auckland, New Zealand
- Peru (3):
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 1702), Lima
  - Oncosalud ( Site 1701), Lima
  - Hospital Militar Central Luis Arias Schereiber ( Site 1700), Lima
- Poland (5):
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością MEDIC-R Sp.k ( Site 0805), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 0801), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Układu Moczowego ( Site 0800), Warsaw, Masovian Voivodeship
  - Oddzial Onkologii Klinicznej z Pododdzialem Chemioterapii Jednodniowej ( Site 0802), Koszalin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 0806), Kielce, Świętokrzyskie Voivodeship
- South Korea (3):
  - Korea University Anam Hospital ( Site 2002), Seoul
  - Seoul National University Hospital-Urology ( Site 2000), Seoul
  - Samsung Medical Center-Urology ( Site 2001), Seoul
- Spain (5):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 1006), Badalona, Barcelona
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 1003), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 1005), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 1002), Barcelona
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 1001), Seville
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna ( Site 1101), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 1102), Uppsala, Uppsala County
- Turkey (Türkiye) (7):
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1200), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1204), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1201), Ankara
  - Koc Universitesi Hastanesi ( Site 1206), Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Baki-Istanbul Bakirkoy Sadi Konuk Training ( Site 1205), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1202), Istanbul
  - Ege Universitesi Hastanesi-Medical Oncology ( Site 1203), Izmir
- United Kingdom (5):
  - Torbay Hospital ( Site 1303), Torquay, Devon
  - Royal Free Hospital ( Site 1300), London, England
  - Gartnavel General Hospital-Clinical Trials Unit ( Site 1301), Glasgow, Glasgow City
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 1302), London, London, City of
  - The Christie NHS Foundation Trust ( Site 1306), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26155&tenant=MT_MSD_9011